CLINICAL TRIAL: NCT02576951
Title: Tolerability, Pharmacokinetics and Pharmacodynamics of LY2951742 in Healthy Subjects Following a Subcutaneous Administration of a Lyophilized Formulation or a Solution Formulation
Brief Title: A Study of Galcanezumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16084; I5Q-MC-CGAO (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-10-14; First posted 2015-10-15 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-02

CONDITIONS: Healthy
MeSH Terms: interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Galcanezumab Solution Formulation-Part A (Experimental): Galcanezumab solution formulation in a prefilled syringe given SC once.
  Interventions: Drug: Galcanezumab
- Placebo-Part A (Placebo Comparator): Placebo in a prefilled syringe given SC once.
  Interventions: Drug: Placebo
- Galcanezumab Lyophilized Formulation-Part B (Experimental): Galcanezumab lyophilized (freeze dried) formulation given SC once.
  Interventions: Drug: Galcanezumab
- Galcanezumab Solution Formulation-Part B (Experimental): Galcanezumab solution formulation in a prefilled syringe given SC once.
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
  Arms: Galcanezumab Lyophilized Formulation-Part B; Galcanezumab Solution Formulation-Part A; Galcanezumab Solution Formulation-Part B
Drug: Placebo — Administered SC
  Arms: Placebo-Part A

SUMMARY:
The purposes of this study are:

* To evaluate tolerability of the Galcanezumab solution injectable formulation (Part A)
* To measure how much of the Galcanezumab lyophilized (freeze dried) injectable formulation is absorbed into the blood stream and how long it takes the body to get rid of it compared to the Galcanezumab solution injectable formulation after a single injection under the skin (subcutaneous [SC]) (Part B).

Information about any side effects that may occur will also be collected. Each part of the study will last about six months. Participants may only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy participants
* Have a body mass index of 19.0 to 35.0 kilograms per meter square (kg/m²), inclusive

Exclusion Criteria:

- Currently smoke in excess of 5 cigarettes/day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2016-09-03 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

REFERENCES:
- [Derived] Kielbasa W, Quinlan T. Population Pharmacokinetics of Galcanezumab, an Anti-CGRP Antibody, Following Subcutaneous Dosing to Healthy Individuals and Patients With Migraine. J Clin Pharmacol. 2020 Feb;60(2):229-239. doi: 10.1002/jcph.1511. Epub 2019 Sep 4. PMID 31482569

RESULTS

PARTICIPANT FLOW:
Groups:
- 240 mg Galcanezumab Solution - Part A: Participants received 240 milligram (mg) Galcanezumab as a solution formulation by subcutaneous injection.
- Placebo - Part A: Participants received placebo by subcutaneous injection.
- 300 mg Galcanezumab Lyophilized - Part B: Participants received 300 mg Galcanezumab as a lyophilized formulation by subcutaneous injection.
- 300 mg Galcanezumab Solution - Part B: Participants received 300 mg Galcanezumab as a solution formulation by subcutaneous injection
Period: Overall Study
Arm/Group | 240 mg Galcanezumab Solution - Part A | Placebo - Part A | 300 mg Galcanezumab Lyophilized - Part B | 300 mg Galcanezumab Solution - Part B
Started | 15 | 3 | 80 | 80
Received at Least One Dose of Study Drug | 15 | 3 | 80 | 80
Completed | 14 | 3 | 78 | 75
Not Completed | 1 | 0 | 2 | 5
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 240 mg Galcanezumab Solution - Part A: Participants received 240 mg Galcanezumab as a solution formulation by subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | 240 mg Galcanezumab Solution - Part A | Placebo - Part A | 300 mg Galcanezumab Lyophilized - Part B | 300 mg Galcanezumab Solution - Part B | Total
Number analyzed (Participants) | 15 | 3 | 80 | 80 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12.1) | 45.7 (14.5) | 38.5 (11.4) | 40.6 (12.8) | 40.5 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 36 | 38 | 86
  Male | 6 | 0 | 44 | 42 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 43 | 36 | 85
  White | 8 | 2 | 30 | 34 | 74
  More than one race | 1 | 0 | 4 | 8 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 3 | 80 | 80 | 178
Basal Metabolic Index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter] | 26.27 (3.86) | 30.67 (4.32) | 27.57 (4.14) | 27.55 (3.97) | 27.56 (4.04)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With an Injection Site Adverse Event
Description: If an injection site reaction is present, it will be fully characterized (including erythema, induration, pain, itching). A summary of other nonserious adverse event (AE), and all serious adverse events (SAE), regardless of causality, is located in the reported adverse events section.
Time Frame: Part A: Predose through 48 hours post dose
Population: All randomized participants who received at least one dose of study drug in Part A and had at least one post dose safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- 240 mg Galcanezumab - Part A: Participants received 240 mg Galcanezumab as a solution formulation by subcutaneous injection.
Arm/Group | 240 mg Galcanezumab - Part A | Placebo - Part A
Number analyzed (Participants) | 15 | 3
Participants | 3 | 0

2. Primary Outcome: Part B: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) From Time Zero to Infinity of Galcanezumab
Description: Part B: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) from Time Zero to Infinity of Galcanezumab.
Time Frame: Part B: Predose,8,24,48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688,3360 hours post dose
Population: All randomized participants who received at least one dose of study drug in Part B and had evaluable AUC zero to infinity PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram per milliliter(day*μg/mL)
Groups:
- 300mg Galcanezumab Solution - Part B: Participants received 300 mg Galcanezumab as a solution formulation by subcutaneous injection.
Arm/Group | 300mg Galcanezumab Solution - Part B | 300 mg Galcanezumab Lyophilized - Part B
Number analyzed (Participants) | 78 | 79
day*microgram per milliliter(day*μg/mL) | 1490 (31) | 1670 (32)

3. Primary Outcome: Part B: Pharmacokinetics: Maximum Concentration (Cmax) of Galcanezumab
Description: Part B: Pharmacokinetics: Maximum Concentration (Cmax) of Galcanezumab.
Time Frame: Part B: Predose,8,24,48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688,3360 hours post dose
Population: All randomized participants who received at least one dose of study drug in part B and had evaluable Cmax PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (μg/mL)
Arm/Group | 300 mg Galcanezumab Solution - Part B | 300 mg Galcanezumab Lyophilized - Part B
Number analyzed (Participants) | 78 | 79
Microgram per milliliter (μg/mL) | 38 (30) | 42.4 (28)

4. Secondary Outcome: Part A: Pharmacodynamics (PD): Time to Maximum Concentration (Tmax) of Plasma Calcitonin Gene Related Peptide (CGRP)
Description: Part A: Pharmacodynamics (PD): Time to maximum concentration (tmax) of Plasma Calcitonin Gene Related Peptide (CGRP).
Time Frame: Part A: Predose,8,24,48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688,3360 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable plasma Tmax CGRP data in Part A.
Measure: Median (Full Range); unit: Days
Arm/Group | 240 mg Galcanezumab - Part A
Number analyzed (Participants) | 14
Days | 56.01 [28.04 to 112.01]

5. Secondary Outcome: Part A: Pharmacodynamics (PD): Area Under the Concentration Versus Time Curve From Time Zero to Tlast (AUC [0 to Tlast]) of Plasma Calcitonin Gene Related Peptide (CGRP)
Description: Part A: Pharmacodynamics (PD): Area Under the Concentration Versus Time Curve From Time Zero to Tlast (AUC [0 to Tlast]) of Plasma Calcitonin Gene Related Peptide (CGRP).
Time Frame: Part A: Predose,8,24,48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688,3360 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable plasma AUC CGRP data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Groups:
- 240 mg Galcanezumab - Part A: Participants received 240mg Galcanezumab as a solution formulation by subcutaneous injection.
Arm/Group | 240 mg Galcanezumab - Part A
Number analyzed (Participants) | 14
day*ng/mL | 231 (48)

6. Secondary Outcome: Part A: Pharmacodynamics (PD): Maximum Concentration (Cmax) of Plasma CGRP
Description: Part A: Pharmacodynamics (PD): Maximum Concentration (Cmax) of Plasma CGRP.
Time Frame: Part A: Predose,8,24,48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688,3360 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable plasma Cmax CGRP data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 240 mg Galcanezumab - Part A
Number analyzed (Participants) | 14
ng/mL | 2.64 (34)

7. Secondary Outcome: Part B: Pharmacodynamics (PD): Time to Maximum Concentration (Tmax) of Plasma Calcitonin Gene Related Peptide (CGRP)
Description: Part B: Pharmacodynamics (PD): Time to maximum concentration (tmax) of Plasma Calcitonin Gene Related Peptide (CGRP).
Time Frame: Part B: Predose, 8,24,48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688,3360 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable plasma Tmax CGRP data in Part B.
Measure: Median (Full Range); unit: Days
Arm/Group | 300 mg Galcanezumab Solution - Part B | 300 mg Galcanezumab Lyophilized - Part B
Number analyzed (Participants) | 78 | 79
Days | 41.93 [20.93 to 84.03] | 41.95 [13.92 to 83.95]

8. Secondary Outcome: Part B: Pharmacodynamics (PD): Area Under the Concentration Versus Time Curve From Time Zero to Tlast (AUC[0-tlast]) of Plasma Calcitonin Gene Related Peptide (CGRP)
Description: Part B: Pharmacodynamics (PD): Area Under the Concentration Versus Time Curve from time zero to tlast (AUC[0-tlast]) of Plasma Calcitonin Gene Related Peptide (CGRP).
Time Frame: Part B: Predose,8,24,48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688,3360 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable plasma AUC zero to tlast CGRP data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | 300 mg Galcanezumab Solution - Part B | 300 mg Galcanezumab Lyophilized - Part B
Number analyzed (Participants) | 75 | 78
day*ng/mL | 169 (50) | 192 (50)

9. Secondary Outcome: Part B: Pharmacodynamics (PD): Maximum Concentration (Cmax) of Plasma CGRP
Description: Part B: Pharmacodynamics (PD): Maximum Concentration (Cmax) of Plasma CGRP.
Time Frame: Part B: Predose,8,24,48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688,3360 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable plasma Cmax CGRP data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 300 mg Galcanezumab Solution - Part B | 300 mg Galcanezumab Lyophilized - Part B
Number analyzed (Participants) | 78 | 79
ng/mL | 2.19 (36) | 2.38 (34)

ADVERSE EVENTS:
Time Frame: Up to 20 Weeks
Description: All randomized participants.
Groups:
- Galcanezumab 240 mg - Part A: Participants received 240 mg Galcanezumab as a solution formulation by subcutaneous injection.
- Galcanezumab 300 mg Lyophilized - Part B: Participants received 300 mg Galcanezumab as a lyophilized formulation by subcutaneous injection.
- Galcanezumab 300 mg Solution - Part B: Participants received 300 mg Galcanezumab as a solution formulation by subcutaneous injection.
Arm/Group | Galcanezumab 240 mg - Part A | Placebo - Part A | Galcanezumab 300 mg Lyophilized - Part B | Galcanezumab 300 mg Solution - Part B
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/3 | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/3 | 1/80 | 0/80
Other Adverse Events (participants affected / at risk) | 7/15 | 1/3 | 25/80 | 20/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galcanezumab 240 mg - Part A (N=15) | Placebo - Part A (N=3) | Galcanezumab 300 mg Lyophilized - Part B (N=80) | Galcanezumab 300 mg Solution - Part B (N=80)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galcanezumab 240 mg - Part A (N=15) | Placebo - Part A (N=3) | Galcanezumab 300 mg Lyophilized - Part B (N=80) | Galcanezumab 300 mg Solution - Part B (N=80)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (4)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biopsy breast (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Physical breast examination abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other